CLINICAL TRIAL: NCT02585778
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Alirocumab in Insulin Treated Patients With Type 1 or Type 2 Diabetes and With Hypercholesterolemia at High Cardiovascular Risk Not Adequately Controlled on Maximally Tolerated LDL-C Lowering Therapy
Brief Title: Efficacy and Safety of Alirocumab Versus Placebo on Top of Maximally Tolerated Lipid Lowering Therapy in Patients With Hypercholesterolemia Who Have Type 1 or Type 2 Diabetes and Are Treated With Insulin (ODYSSEY DM - Insulin)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LPS14355; 2015-000799-92 (EudraCT Number); U1111-1172-4772 (Other: UTN)
Record Dates: First submitted 2015-10-22; First posted 2015-10-23 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-04

CONDITIONS: Hypercholesterolaemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab; Hypoglycemic Agents

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alirocumab 75 mg Q2W/Up to 150 mg Q2W (Experimental): Alirocumab 75 mg subcutaneous (SC) injection every 2 weeks (Q2W) added to stable, maximally tolerated dose of statin therapy with or without other lipid-modifying therapy (LMT), insulin alone or with other antihyperglycemic drugs for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when LDL-C levels ≥70 mg/dL (1.81 mmol/L) at Week 8.
  Interventions: Drug: Alirocumab; Drug: Lipid-Modifying Therapy (LMT); Drug: Antihyperglycemic Drug
- Placebo Q2W (Placebo Comparator): Placebo (for alirocumab) SC injection Q2W added to stable, maximally tolerated dose of statin therapy with or without other LMT, insulin alone or with other antihyperglycemic drugs for 24 weeks.
  Interventions: Drug: Placebo; Drug: Lipid-Modifying Therapy (LMT); Drug: Antihyperglycemic Drug

INTERVENTIONS:
Drug: Alirocumab — Solution for injection, one subcutaneous injection in the abdomen, thigh, or outer area of upper arm with a disposable auto-injector.
  Other Names: Praluent; SAR236553; REGN727
  Arms: Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Drug: Placebo — Solution for injection, one subcutaneous injection in the abdomen, thigh, or outer area of upper arm with a disposable auto-injector.
  Arms: Placebo Q2W
Drug: Lipid-Modifying Therapy (LMT) — Statins at stable, maximally tolerated dose with or without other LMT as clinically indicated.
Drug: Antihyperglycemic Drug — Insulin (injectable or inhaled) alone or with other antihyperglycemic drugs as clinically indicated.

SUMMARY:
Primary Objectives:

* To demonstrate the superiority of alirocumab in comparison with placebo in the reduction of calculated low-density lipoprotein cholesterol (LDL-C) in participants with diabetes treated with insulin and with hypercholesterolemia at high cardiovascular risk not adequately controlled on maximally tolerated LDL-C lowering therapy.
* To evaluate the safety and tolerability of alirocumab in participants with diabetes treated with insulin.

Secondary Objective:

To demonstrate that alirocumab was superior in comparison to placebo in its effects on other lipid parameters (i.e., measured LDL-C, non-high-density lipoprotein cholesterol [non-HDL-C], apolipoprotein B [Apo B], total cholesterol [TC], lipoprotein a [Lp(a)], high density lipoprotein cholesterol [HDL-C], triglyceride [TG] levels, triglyceride rich lipoproteins [TGRL], apolipoprotein A-1 [Apo A-1], apolipoprotein C-III [Apo C-III], and LDL particle number and size).

DETAILED DESCRIPTION:
The maximum study duration was approximately 9 months per participant, including a 6 month treatment period, a screening period of up to 3 weeks, and an 8 week safety observation period.

ELIGIBILITY:
Inclusion criteria:

* Participants diagnosed with Type 1 or Type 2 diabetes at least one year prior to the screening visit (Week -3).
* Signed written informed consent
* Participants with type 1 or type 2 diabetes treated with insulin whose LDL-C levels were not adequately controlled with maximally tolerated lipid-modifying therapy
* LDL-C of 70 mg/dL or greater
* 18 years of age or more
* Glycosylated hemoglobin (HbA1c) less than 10%
* History of cardiovascular disease (including coronary heart disease [CHD] and/or CHD risk equivalents) and/or at least one additional cardiovascular risk factor

Exclusion criteria:

* Not on a stable dose of statin or other lipid modifying therapy for at least 4 weeks prior to screening or from screening to randomization, unless statin intolerant
* Triglycerides >400 mg/dL
* Estimated glomerular filtration rate (eGFR) <15 mL/min/1.73 m² according to the Modification of Diet in Renal Disease (MDRD) equation
* Currently received or planned to receive renal replacement therapy (for example, hemodialysis)
* Change in weight of more than 5 kilograms within the prior 2 months
* Not on a stable dose/regimen of insulin or other antidiabetic drugs for the past 3 months or planned to intensify insulin regimen during the study
* Not treated with insulin for at least 6 months
* Planned to start new lipid modifying therapy or change dose of current lipid modifying therapy during the study
* Body mass index (BMI) >45 kg/m² or planned to undergo bariatric surgery, weight loss program, or initiate weight loss drugs during the study
* History of recent decompensation of diabetes within the prior 2 months (for example, diabetic ketoacidosis)

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2015-10-23 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2017-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (110):
- United States (29):
  - Investigational Site Number 840020, Encino, California
  - Investigational Site Number 840002, Fresno, California
  - Investigational Site Number 840029, Oakland, California
  - Investigational Site Number 840027, Loveland, Colorado
  - Investigational Site Number 840026, Atlantis, Florida
  - Investigational Site Number 840006, Bradenton, Florida
  - Investigational Site Number 840023, Jacksonville, Florida
  - Investigational Site Number 840028, Palm Harbor, Florida
  - Investigational Site Number 840022, Ponte Vedra Beach, Florida
  - Investigational Site Number 840021, Roswell, Georgia
  - Investigational Site Number 840007, Springfield, Illinois
  - Investigational Site Number 840011, Indianapolis, Indiana
  - Investigational Site Number 840015, Valparaiso, Indiana
  - Investigational Site Number 840010, Des Moines, Iowa
  - Investigational Site Number 840005, Louisville, Kentucky
  - Investigational Site Number 840018, Auburn, Maine
  - Investigational Site Number 840013, Hyattsville, Maryland
  - Investigational Site Number 840016, Rockville, Maryland
  - Investigational Site Number 840004, Minneapolis, Minnesota
  - Investigational Site Number 840012, Jamaica, New York
  - Investigational Site Number 840014, Maumee, Ohio
  - Investigational Site Number 840009, Greer, South Carolina
  - Investigational Site Number 840024, Chattanooga, Tennessee
  - Investigational Site Number 840001, Austin, Texas
  - Investigational Site Number 840003, Dallas, Texas
  - Investigational Site Number 840019, Dallas, Texas
  - Investigational Site Number 840025, Houston, Texas
  - Investigational Site Number 840017, Ogden, Utah
  - Investigational Site Number 840008, Salt Lake City, Utah
- Austria (5):
  - Investigational Site Number 040002, Innsbruck
  - Investigational Site Number 040005, Linz
  - Investigational Site Number 040003, Salzburg
  - Investigational Site Number 040004, Salzburg
  - Investigational Site Number 040001, Vienna
- Belgium (3):
  - Investigational Site Number 056002, Edegem
  - Investigational Site Number 056003, Haine-Saint-Paul
  - Investigational Site Number 056001, Leuven
- France (9):
  - Investigational Site Number 250-008, Besançon
  - Investigational Site Number 250-005, Corbeil-Essonnes
  - Investigational Site Number 250-004, La Rochelle
  - Investigational Site Number 250-003, Le Creusot
  - Investigational Site Number 250-009, Mulhouse
  - Investigational Site Number 250-002, Nantes
  - Investigational Site Number 250-007, Paris
  - Investigational Site Number 250-006, Strasbourg
  - Investigational Site Number 250-001, Toulouse
- Germany (18):
  - Investigational Site Number 276015, Aschaffenburg
  - Investigational Site Number 276002, Berlin
  - Investigational Site Number 276011, Dortmund
  - Investigational Site Number 276019, Dresden
  - Investigational Site Number 276014, Dresden
  - Investigational Site Number 276009, Dresden
  - Investigational Site Number 276021, Hamburg
  - Investigational Site Number 276018, Hamburg
  - Investigational Site Number 276005, Heidelberg
  - Investigational Site Number 276013, Lüneburg
  - Investigational Site Number 276022, Magdeburg
  - Investigational Site Number 276008, Neumünster
  - Investigational Site Number 276017, Neuwied
  - Investigational Site Number 276004, Oldenburg
  - Investigational Site Number 276003, Pirna
  - Investigational Site Number 276006, Riesa
  - Investigational Site Number 276010, Saarlouis
  - Investigational Site Number 276016, Sulzbach-Rosenberg
- Italy (12):
  - Investigational Site Number 380004, Catania
  - Investigational Site Number 380003, Catanzaro
  - Investigational Site Number 380011, Como
  - Investigational Site Number 380006, Milan
  - Investigational Site Number 380007, Milan
  - Investigational Site Number 380005, Moncalieri
  - Investigational Site Number 380009, Napoli
  - Investigational Site Number 380008, Padua
  - Investigational Site Number 380002, Palermo
  - Investigational Site Number 380001, Pisa
  - Investigational Site Number 380010, Roma
  - Investigational Site Number 380012, Verona
- Netherlands (5):
  - Investigational Site Number 528002, Apeldoorn
  - Investigational Site Number 528005, Groningen
  - Investigational Site Number 528003, Hoogeveen
  - Investigational Site Number 528001, Rotterdam
  - Investigational Site Number 528004, Utrecht
- Spain (14):
  - Investigational Site Number 724007, Badalona
  - Investigational Site Number 724001, Barcelona
  - Investigational Site Number 724006, Ferrol
  - Investigational Site Number 724013, Granada
  - Investigational Site Number 724005, Madrid
  - Investigational Site Number 724004, Madrid
  - Investigational Site Number 724011, Majadahonda
  - Investigational Site Number 724008, Málaga
  - Investigational Site Number 724014, Oviedo
  - Investigational Site Number 724009, Palma de Mallorca
  - Investigational Site Number 724002, Pamplona
  - Investigational Site Number 724010, Sant Joan Despí
  - Investigational Site Number 724012, Segovia
  - Investigational Site Number 724003, Seville
- Switzerland (2):
  - Investigational Site Number 756001, Olten
  - Investigational Site Number 756003, Sankt Gallen
- United Kingdom (13):
  - Investigational Site Number 826010, Airdrie
  - Investigational Site Number 826011, Bath
  - Investigational Site Number 826009, Bournemouth
  - Investigational Site Number 826005, Bradford
  - Investigational Site Number 826004, Bristol
  - Investigational Site Number 826001, Burton-on-Trent
  - Investigational Site Number 826015, Durham
  - Investigational Site Number 826012, High Wycombe
  - Investigational Site Number 826007, Manchester
  - Investigational Site Number 826006, Peterborough
  - Investigational Site Number 826003, Southampton
  - Investigational Site Number 826008, Truro
  - Investigational Site Number 826002, Welwyn Garden City

REFERENCES:
- [Derived] Schmidt AF, Carter JL, Pearce LS, Wilkins JT, Overington JP, Hingorani AD, Casas JP. PCSK9 monoclonal antibodies for the primary and secondary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2020 Oct 20;10(10):CD011748. doi: 10.1002/14651858.CD011748.pub3. PMID 33078867
- [Derived] Ray KK, Del Prato S, Muller-Wieland D, Cariou B, Colhoun HM, Tinahones FJ, Domenger C, Letierce A, Mandel J, Samuel R, Bujas-Bobanovic M, Leiter LA. Alirocumab therapy in individuals with type 2 diabetes mellitus and atherosclerotic cardiovascular disease: analysis of the ODYSSEY DM-DYSLIPIDEMIA and DM-INSULIN studies. Cardiovasc Diabetol. 2019 Nov 9;18(1):149. doi: 10.1186/s12933-019-0951-9. PMID 31706300
- [Derived] Leiter LA, Cariou B, Muller-Wieland D, Colhoun HM, Del Prato S, Tinahones FJ, Ray KK, Bujas-Bobanovic M, Domenger C, Mandel J, Samuel R, Henry RR. Efficacy and safety of alirocumab in insulin-treated individuals with type 1 or type 2 diabetes and high cardiovascular risk: The ODYSSEY DM-INSULIN randomized trial. Diabetes Obes Metab. 2017 Dec;19(12):1781-1792. doi: 10.1111/dom.13114. Epub 2017 Oct 10. PMID 28905478

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 103 sites in 10 countries. Of these, 97 active sites randomized at least 1 participant. Overall 796 participants were screened between October 2015 and August 2016, of whom 279 were screen failures. Screen failures were mainly due to exclusion criteria met or inclusion criteria not met.
Pre-assignment Details: Randomization was stratified by diabetes type (Type 1 diabetes mellitus [T1DM] versus Type 2 diabetes mellitus [T2DM]). Assignment to treatment arms was done centrally using an Interactive Voice/Web Response System in a 2:1 ratio (Alirocumab:Placebo). A total of 517 participants were randomized. Baseline and efficacy data were analyzed per stratum.
Groups:
- Alirocumab 75 mg Q2W/Up to 150 mg Q2W: Alirocumab 75 mg subcutaneous (SC) injection every 2 weeks (Q2W) added to stable, maximally tolerated dose of statin therapy with or without other lipid-modifying therapy (LMT), insulin alone or with other antihyperglycemic drugs for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when low-density lipoprotein cholesterol (LDL-C) levels ≥70 mg/dL (1.81 mmol/L) at Week 8.
Period: Overall Study
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Placebo Q2W
Started | 345 (Randomized) | 172 (Randomized)
Treated (Safety Population) | 344 | 170
ITT Population | 336 | 167
mITT Population | 333 | 164
T1DM Participants (Randomized stratum: T1DM) | 51 | 25
T2DM Participants (Randomized stratum: T2DM) | 294 | 147
Completed (Completed = treatment completion) | 312 | 157
Not Completed | 33 | 15
Not completed — Adverse Event | 17 | 4
Not completed — Participant did not wish to continue | 9 | 4
Not completed — Poor compliance to study protocol | 0 | 2
Not completed — Death | 0 | 1
Not completed — Randomized but not treated | 1 | 2
Not completed — Other than specified above | 6 | 2

BASELINE CHARACTERISTICS:
Population: Baseline population included all randomized participants.
Groups:
- Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants; Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants: Alirocumab 75 mg SC injection Q2W added to stable, maximally tolerated dose of statin therapy with or without other LMT, insulin alone or with other antihyperglycemic drugs for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when LDL-C levels ≥70 mg/dL (1.81 mmol/L) at Week 8.
- Placebo Q2W: T1DM Participants; Placebo Q2W: T2DM Participants: Placebo (for alirocumab) SC injection Q2W added to stable, maximally tolerated dose of statin therapy with or without other LMT, insulin alone or with other antihyperglycemic drugs for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants | Total
Number analyzed (Participants) | 51 | 25 | 294 | 147 | 517
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (10.1) | 58.5 (7.8) | 63.9 (8.9) | 64.0 (9.4) | 62.8 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 8 | 133 | 69 | 232
  Male | 29 | 17 | 161 | 78 | 285
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 13 | 8 | 22
  Not Hispanic or Latino | 50 | 25 | 280 | 138 | 493
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 50 | 24 | 259 | 135 | 468
  Black | 1 | 0 | 27 | 7 | 35
  Asian/Oriental | 0 | 0 | 7 | 3 | 10
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Other | 0 | 1 | 1 | 2 | 4
Calculated LDL-C in mg/dL [Mean (Standard Deviation); unit: mg/dL] — Calculated LDL-C in mg/dL from Friedewald formula (LDL cholesterol = Total cholesterol - high density lipoprotein [HDL] cholesterol - [Triglyceride/5]).
  mg/dL | 126.4 (58.2) | 110.2 (31.2) | 110.8 (36.5) | 109.6 (39.1) | 112.0 (39.8)
Calculated LDL-C in mmol/L [Mean (Standard Deviation); unit: mmol/L] — Calculated LDL-C in mmol/L from Friedewald formula (LDL cholesterol = Total cholesterol - HDL cholesterol - [Triglyceride/2.2]).
  mmol/L | 3.273 (1.506) | 2.853 (0.807) | 2.871 (0.944) | 2.838 (1.013) | 2.900 (1.031)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - Intent-to-treat (ITT) Analysis
Description: Adjusted Least-squares (LS) means and standard errors at Week 24 were obtained from a mixed-effect model with repeated measures (MMRM) to account for missing data. All available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment were used in the model (ITT analysis).
Time Frame: From Baseline to Week 24
Population: ITT population: all randomized participants with one baseline and at least one post-baseline calculated LDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 49 | 25 | 287 | 142
percent change | -51.8 (3.7) | -3.9 (5.3) | -48.2 (1.6) | 0.8 (2.2)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants vs Placebo Q2W: T1DM Participants; Alirocumab group was compared to placebo group using an appropriate contrast statement; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -47.8, 95% CI 2-sided [-60.7 to -35.0] — Alirocumab vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants vs Placebo Q2W: T2DM Participants; Alirocumab group was compared to placebo group using an appropriate contrast statement; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -49.0, 95% CI 2-sided [-54.4 to -43.6] — Alirocumab vs. Placebo

2. Primary Outcome: Percentage of Participants Who Experienced Treatment-Emergent Adverse Events (AEs)
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'treatment-emergent period' (the time from the first dose of study drug up to the last dose of study drug +70 days).
Time Frame: From Baseline up to 10 weeks after last study drug administration (maximum of 32 weeks)
Population: Safety population: all randomized participants who received at least one dose or part of a dose of a study drug (treated).
Measure: Number; unit: percentage of participants
Groups:
- Alirocumab 75 mg Q2W/Up to 150 mg Q2W: Alirocumab 75 mg SC injection Q2W added to stable, maximally tolerated dose of statin therapy with or without other LMT, insulin alone or with other antihyperglycemic drugs for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when LDL-C levels ≥70 mg/dL (1.81 mmol/L) at Week 8.
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Placebo Q2W
Number analyzed (Participants) | 344 | 170
percentage of participants
  Any AE | 64.5 | 64.1
  Any Serious AE | 9.0 | 9.4
  Any AE leading to death | 0 | 0.6
  Any AE leading to treatment discontinuation | 4.9 | 2.4

3. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 were obtained from MMRM model including available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 24
Population: Modified ITT population (mITT): all randomized and treated participants with one baseline and at least one post-baseline calculated LDL-C value on-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 49 | 24 | 284 | 140
percent change | -53.8 (3.7) | -3.2 (5.3) | -50.9 (1.6) | 0.7 (2.2)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants vs Placebo Q2W: T1DM Participants; A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 0.05 level. Hierarchical testing procedure was followed for T1DM and T2DM participants separately; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -50.6, 95% CI 2-sided [-63.4 to -37.9] — Alirocumab vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants vs Placebo Q2W: T2DM Participants; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant in relevant diabetes stratum); Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -51.6, 95% CI 2-sided [-56.9 to -46.4] — Alirocumab vs. Placebo

4. Secondary Outcome: Percent Change From Baseline in Measured LDL-C at Week 24 - ITT Analysis
Description: Measured LDL-C values via beta quantification method. Adjusted LS means and standard errors at Week 24 from MMRM model including available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline measured LDL-C value on- or off-treatment (Measured LDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 47 | 22 | 277 | 139
percent change | -49.4 (3.7) | -1.1 (5.4) | -43.3 (1.6) | 2.4 (2.2)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants vs Placebo Q2W: T1DM Participants; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -48.4, 95% CI 2-sided [-61.2 to -35.5] — Alirocumab vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants vs Placebo Q2W: T2DM Participants; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -45.7, 95% CI 2-sided [-50.9 to -40.4] — Alirocumab vs. Placebo

5. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline calculated LDL-C value on- or off-treatment at Week 12 (ITT population at Week 12).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 49 | 25 | 284 | 140
percent change | -49.4 (3.5) | -4.5 (5.0) | -48.8 (1.4) | 1.4 (2.1)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants vs Placebo Q2W: T1DM Participants; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -44.8, 95% CI 2-sided [-56.9 to -32.8] — Alirocumab vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants vs Placebo Q2W: T2DM Participants; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -50.2, 95% CI 2-sided [-55.2 to -45.3] — Alirocumab vs. Placebo

6. Secondary Outcome: Percent Change From Baseline in Measured LDL-C at Week 12 - ITT Analysis
Description: Measured LDL-C values via beta quantification method. Adjusted LS means and standard errors at Week 12 from MMRM model including available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline measured LDL-C value on- or off-treatment at Week 12 (Measured LDL-C ITT population at Week 12).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 45 | 22 | 275 | 136
percent change | -46.7 (3.6) | -4.0 (5.1) | -44.8 (1.4) | -0.8 (2.0)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants vs Placebo Q2W: T1DM Participants; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -42.7, 95% CI 2-sided [-54.9 to -30.5] — Alirocumab vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants vs Placebo Q2W: T2DM Participants; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -44.1, 95% CI 2-sided [-49.0 to -39.2] — Alirocumab vs. Placebo

7. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 24 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline non-HDL-C value on- or off-treatment (non-HDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 49 | 25 | 287 | 142
percent change | -45.9 (3.3) | -3.2 (4.8) | -37.9 (1.4) | 0.7 (2.0)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants vs Placebo Q2W: T1DM Participants; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -42.7, 95% CI 2-sided [-54.2 to -31.3] — Alirocumab vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants vs Placebo Q2W: T2DM Participants; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -38.7, 95% CI 2-sided [-43.4 to -33.9] — Alirocumab vs. Placebo

8. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (Apo-B) at Week 24 - ITT Analysis
Description: as for outcome 7
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline Apo B value on- or off-treatment (Apo B ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 47 | 22 | 279 | 140
percent change | -39.4 (3.0) | -0.4 (4.3) | -33.4 (1.3) | 3.3 (1.7)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants vs Placebo Q2W: T1DM Participants; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -39.0, 95% CI 2-sided [-49.4 to -28.7] — Alirocumab vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants vs Placebo Q2W: T2DM Participants; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -36.7, 95% CI 2-sided [-40.9 to -32.5] — Alirocumab vs. Placebo

9. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Total-C) at Week 24 - ITT Analysis
Description: as for outcome 7
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline total-C value on- or off-treatment (Total-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 49 | 25 | 287 | 142
percent change | -29.9 (2.5) | -0.7 (3.6) | -26.8 (1.0) | 0.8 (1.5)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants vs Placebo Q2W: T1DM Participants; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -29.2, 95% CI 2-sided [-37.8 to -20.7] — Alirocumab vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants vs Placebo Q2W: T2DM Participants; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -27.6, 95% CI 2-sided [-31.2 to -24.1] — Alirocumab vs. Placebo

10. Secondary Outcome: Percentage of Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - On-Treatment Analysis
Description: Adjusted percentages at Week 24 from multiple imputation approach model including available post-baseline data from Week 4 to Week 24 (i.e. up to 21 days after last injection).
Time Frame: Up to Week 24
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 49 | 24 | 284 | 140
percentage of participants | 70.2 | 5.1 | 76.4 | 7.4
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants vs Placebo Q2W: T1DM Participants; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.0001, Regression, Logistic — Threshold for significance at 0.05 level; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 117.0, 95% CI 2-sided [13.1 to 1041.8] — Alirocumab vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants vs Placebo Q2W: T2DM Participants; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.0001, Regression, Logistic — Threshold for significance at 0.05 level; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 84.6, 95% CI 2-sided [36.5 to 196.1] — Alirocumab vs. Placebo

11. Secondary Outcome: Percentage of Participants Reaching Calculated LDL-C <50 mg/dL (1.3 mmol/L) at Week 24 - On-Treatment Analysis
Description: Adjusted percentages at Week 24 from last observation carried forward (LOCF) approach (for T1DM participants) and multiple imputation approach model (for T2DM participants) including available post-baseline data from Week 4 to Week 24 (i.e. up to 21 days after last injection). The maximum likelihood estimate did not exist as response rate was zero in a treatment group of T1DM participants.
Time Frame: Up to Week 24
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 49 | 24 | 284 | 140
percentage of participants | 55.1 | 0 | 50.7 | 2.7
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants vs Placebo Q2W: T2DM Participants; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority; p < 0.0001, Regression, Logistic — Threshold for significance at 0.05 level; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 52.9, 95% CI 2-sided [16.6 to 168.3] — Alirocumab vs. Placebo

12. Secondary Outcome: Percentage of Participants Reaching Calculated Non-HDL-C <100 mg/dL at Week 24 - On-Treatment Analysis
Description: as for outcome 10
Time Frame: Up to Week 24
Population: Participants of the mITT population with one baseline and at least one post-baseline Non-HDL-C value on-treatment (Non-HDL-C mITT population).
Measure: Number; unit: percentage of participants
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 49 | 24 | 284 | 140
percentage of participants | 79.0 | 22.9 | 70.9 | 13.8
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants vs Placebo Q2W: T1DM Participants; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.0001, Regression, Logistic — Threshold for significance at 0.05 level; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 33.2, 95% CI 2-sided [8.0 to 137.4] — Alirocumab vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants vs Placebo Q2W: T2DM Participants; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.0001, Regression, Logistic — Threshold for significance at 0.05 level; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 27.1, 95% CI 2-sided [14.2 to 51.5] — Alirocumab vs. Placebo

13. Secondary Outcome: Percentage of Participants Reaching Calculated Non-HDL-C <80 mg/dL at Week 24 - On-Treatment Analysis
Description: Adjusted percentages at Week 24 from multiple imputation approach including available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection).
Time Frame: Up to Week 24
Population: Non-HDL-C mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 49 | 24 | 284 | 140
percentage of participants | 59.6 | 5.3 | 52.3 | 1.7
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants vs Placebo Q2W: T1DM Participants; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.0002, Regression, Logistic — Threshold for significance at 0.05 level; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 55.5, 95% CI 2-sided [6.5 to 473.7] — Alirocumab vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants vs Placebo Q2W: T2DM Participants; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.0001, Regression, Logistic — Threshold for significance at 0.05 level; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 103.3, 95% CI 2-sided [24.6 to 433.1] — Alirocumab vs. Placebo

14. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at Week 24 - ITT Analysis
Description: Adjusted means and standard errors at Week 24 were obtained from multiple imputation approach for handling of missing data followed by robust regression model. All available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment were included in the imputation model.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 49 | 25 | 287 | 142
percent change | -23.0 (3.8) | -4.3 (5.3) | -19.0 (1.6) | -0.5 (2.2)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants vs Placebo Q2W: T1DM Participants; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.0039, Regression, Robust — Threshold for significance at 0.05 level; Multiple imputation approach followed by robust regression model; Adjusted Mean Difference = -18.7, 95% CI 2-sided [-31.4 to -6.0] — Alirocumab vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants vs Placebo Q2W: T2DM Participants; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.0001, Regression, Robust — Threshold for significance at 0.05 level; Multiple imputation approach followed by robust regression model; Adjusted Mean Difference = -18.4, 95% CI 2-sided [-23.7 to -13.2] — Alirocumab vs. Placebo

15. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 24 - ITT Analysis
Description: as for outcome 7
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline HDL-C value on- or off-treatment (HDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 49 | 25 | 287 | 142
percent change | 11.2 (2.4) | 7.3 (3.5) | 8.1 (1.0) | 3.7 (1.4)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants vs Placebo Q2W: T1DM Participants; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.3434, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = 3.9, 95% CI 2-sided [-4.2 to 12.0] — Alirocumab vs. Placebo
Statistical Analysis 2: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants vs Placebo Q2W: T2DM Participants; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.0100, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = 4.4, 95% CI 2-sided [1.1 to 7.7] — Alirocumab vs. Placebo

16. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 24 - ITT Analysis
Description: Adjusted means and standard errors at Week 24 from multiple imputation approach for handling of missing data followed by robust regression model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 49 | 25 | 287 | 142
percent change | -13.6 (4.7) | 1.9 (6.7) | -5.7 (2.0) | 0.0 (2.7)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants vs Placebo Q2W: T2DM Participants; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.0902, Regression, Robust — Threshold for significance at 0.05 level; Multiple imputation approach followed by robust regression model; Adjusted Mean Difference = -5.7, 95% CI 2-sided [-12.3 to 0.9] — Alirocumab vs. Placebo

17. Secondary Outcome: Percent Change From Baseline in LDL-C Particle Number at Week 24 - ITT Analysis
Description: LDL-C particle number was calculated from lipid subfractions by nuclear magnetic resonance (NMR) spectroscopy. Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline LDL-C particle number value on- or off-treatment (LDL-C particle number ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 45 | 22 | 272 | 134
percent change | -44.4 (3.2) | -4.4 (4.6) | -38.3 (1.3) | 1.9 (1.9)

18. Secondary Outcome: Percent Change From Baseline in LDL-C Particle Size at Week 24 - ITT Analysis
Description: LDL-C particle size was calculated from lipid subfractions by NMR spectroscopy. Adjusted LS means and standard errors at Week 24 from MMRM model including available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline LDL-C particle size value on- or off-treatment (LDL-C particle size ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 44 | 22 | 267 | 134
percent change | -2.3 (0.3) | 0.8 (0.5) | -2.8 (0.1) | -0.3 (0.2)

19. Secondary Outcome: Absolute Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Weeks 12 and 24 - ITT Analysis
Description: Absolute change = HbA1c value at specified weeks minus HbA1c value at baseline.
Time Frame: Baseline, Weeks 12 and 24
Population: ITT population. Here, 'Number Analyzed' = participants with available data at the specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 49 | 25 | 287 | 142
percentage of hemoglobin
  Change at Week 12: number analyzed (Participants) | 48 | 22 | 281 | 138
  Change at Week 12 | 0.00 (0.46) | -0.22 (0.39) | -0.04 (0.57) | 0.00 (0.58)
  Change at Week 24: number analyzed (Participants) | 47 | 22 | 261 | 135
  Change at Week 24 | -0.03 (0.60) | -0.23 (0.36) | 0.18 (0.74) | 0.06 (0.66)

20. Secondary Outcome: Absolute Change From Baseline in HbA1c at Weeks 12 and 24 - On-Treatment Analysis
Description: Absolute change = HbA1c value at specified weeks minus HbA1c value at baseline.
Time Frame: Baseline, Weeks 12 and 24
Population: mITT population. Here, 'Number Analyzed' = participants with available data at the specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 49 | 24 | 284 | 140
percentage of hemoglobin
  Change at Week 12: number analyzed (Participants) | 48 | 22 | 275 | 136
  Change at Week 12 | 0.00 (0.46) | -0.22 (0.39) | -0.04 (0.57) | 0.00 (0.59)
  Change at Week 24: number analyzed (Participants) | 43 | 20 | 243 | 129
  Change at Week 24 | -0.05 (0.61) | -0.27 (0.34) | 0.18 (0.74) | 0.06 (0.67)

21. Secondary Outcome: Absolute Change From Baseline in Fasting Plasma Glucose (FPG) at Weeks 12 and 24 - ITT Analysis
Description: Absolute change = FPG value at specified weeks minus FPG value at baseline.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 49 | 25 | 287 | 142
mmol/L
  Change at Week 12: number analyzed (Participants) | 46 | 20 | 278 | 138
  Change at Week 12 | 0.23 (4.44) | 0.45 (4.73) | 0.25 (2.73) | 0.13 (2.73)
  Change at Week 24: number analyzed (Participants) | 46 | 22 | 257 | 135
  Change at Week 24 | 0.52 (5.20) | 0.81 (4.21) | 0.52 (3.43) | 0.55 (2.62)

22. Secondary Outcome: Absolute Change From Baseline in FPG at Weeks 12 and 24 - On-Treatment Analysis
Description: Absolute change = FPG value at specified weeks minus FPG value at baseline.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 49 | 24 | 284 | 140
mmol/L
  Change at Week 12: number analyzed (Participants) | 46 | 20 | 272 | 136
  Change at Week 12 | 0.23 (4.44) | 0.45 (4.73) | 0.22 (2.70) | 0.15 (2.74)
  Change at Week 24: number analyzed (Participants) | 42 | 20 | 240 | 129
  Change at Week 24 | 0.38 (5.24) | 0.71 (4.19) | 0.52 (3.47) | 0.48 (2.53)

23. Secondary Outcome: Absolute Change From Baseline in Total Daily Insulin Dose at Weeks 12 and 24 - ITT Analysis
Description: Absolute change = total daily insulin dose at specified weeks minus baseline value.
Time Frame: Baseline, Weeks 12 and 24
Population: ITT population . Here, 'Number Analyzed' = participants with available data at the specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units (U)
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 49 | 25 | 287 | 142
units (U)
  Change at Week 12: number analyzed (Participants) | 47 | 21 | 279 | 136
  Change at Week 12 | -10.0 (48.7) | -1.3 (9.6) | 0.2 (7.9) | 1.4 (11.4)
  Change at Week 24: number analyzed (Participants) | 48 | 23 | 258 | 130
  Change at Week 24 | -2.2 (11.3) | -0.8 (9.8) | 2.2 (14.8) | 1.6 (11.4)

24. Secondary Outcome: Absolute Change From Baseline in Total Daily Insulin Dose at Weeks 12 and 24 - On-Treatment Analysis
Description: Absolute change = total daily insulin dose at specified weeks minus baseline value.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: units (U)
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 49 | 24 | 284 | 140
units (U)
  Change at Week 12: number analyzed (Participants) | 47 | 21 | 278 | 135
  Change at Week 12 | -10.0 (48.7) | -1.3 (9.6) | 0.2 (7.9) | 1.4 (11.4)
  Change at Week 24: number analyzed (Participants) | 48 | 23 | 257 | 129
  Change at Week 24 | -2.2 (11.3) | -0.8 (9.8) | 1.7 (11.7) | 1.6 (11.5)

25. Secondary Outcome: Absolute Change From Baseline in Insulin Daily Dose/Kg at Weeks 12 and 24 - ITT Analysis
Description: Absolute change = daily insulin dose/kg at specified weeks minus baseline value.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: U/kg
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 49 | 25 | 287 | 142
U/kg
  Change at Week 12: number analyzed (Participants) | 47 | 21 | 279 | 136
  Change at Week 12 | -0.1 (0.5) | 0.0 (0.1) | 0.0 (0.1) | 0.0 (0.1)
  Change at Week 24: number analyzed (Participants) | 48 | 23 | 258 | 130
  Change at Week 24 | 0.0 (0.1) | 0.0 (0.1) | 0.0 (0.2) | 0.0 (0.1)

26. Secondary Outcome: Absolute Change From Baseline in Insulin Daily Dose/Kg at Weeks 12 and 24 - On-Treatment Analysis
Description: Absolute change = daily insulin dose/kg at specified weeks minus baseline value.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: U/kg
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 49 | 24 | 284 | 140
U/kg
  Change at Week 12: number analyzed (Participants) | 47 | 21 | 278 | 135
  Change at Week 12 | -0.1 (0.5) | 0.0 (0.1) | 0.0 (0.1) | 0.0 (0.1)
  Change at Week 24: number analyzed (Participants) | 48 | 23 | 257 | 129
  Change at Week 24 | 0.0 (0.1) | 0.0 (0.1) | 0.0 (0.1) | 0.0 (0.1)

27. Secondary Outcome: Absolute Change From Baseline in Number of Glucose-Lowering Treatments at Weeks 12 and 24 - ITT Analysis
Description: Glucose lowering treatment was calculated for non-insulin treatments as one for each unique treatment received and for insulin treatment as one in total for all participants who have taken one or more treatments. Absolute change = number of glucose-lowering treatments at specified weeks minus baseline value.
Time Frame: Baseline, Weeks 12 and 24
Population: ITT population.
Measure: Mean (Standard Deviation); unit: glucose lowering treatments
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 49 | 25 | 287 | 142
glucose lowering treatments
  Change at Week 12 | 0 (0) | 0 (0) | 0 (0.1) | 0 (0.2)
  Change at Week 24 | 0 (0) | 0 (0) | 0 (0.3) | 0 (0.2)

28. Secondary Outcome: Absolute Change From Baseline in Number of Glucose-Lowering Treatments at Weeks 12 and 24 - On-Treatment Analysis
Description: as for outcome 27
Time Frame: Baseline, Weeks 12 and 24
Population: mITT population.
Measure: Mean (Standard Deviation); unit: glucose lowering treatments
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T1DM Participants | Placebo Q2W: T1DM Participants | Alirocumab 75 mg Q2W/Up to 150 mg Q2W: T2DM Participants | Placebo Q2W: T2DM Participants
Number analyzed (Participants) | 49 | 24 | 284 | 140
glucose lowering treatments
  Change at Week 12 | 0 (0) | 0 (0) | 0 (0.1) | 0 (0.2)
  Change at Week 24 | 0 (0) | 0 (0) | 0 (0.3) | 0 (0.2)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to final visit (Week 32) in the study regardless of seriousness or relationship to study drugs.
Description: Reported AEs and deaths are TEAEs that is AEs that developed/worsened and death that occurred during the 'treatment-emergent period' (the time from the first dose of study drug up to the last dose of study drug +70 days).
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Placebo Q2W
All-Cause Mortality (participants affected / at risk) | 0/344 | 1/170
Serious Adverse Events (participants affected / at risk) | 31/344 | 16/170
Other Adverse Events (participants affected / at risk) | 17/344 | 9/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alirocumab 75 mg Q2W/Up to 150 mg Q2W (N=344) | Placebo Q2W (N=170)
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1
Diabetic foot infection (Infections and infestations) | 1 | 0
Endometritis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2
Pyelonephritis acute (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Pseudoradicular syndrome (Nervous system disorders) | 0 | 1
Radicular syndrome (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alirocumab 75 mg Q2W/Up to 150 mg Q2W (N=344) | Placebo Q2W (N=170)
Nasopharyngitis (Infections and infestations) | 17 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2015-07-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT02585778/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT02585778/SAP_001.pdf